CLINICAL TRIAL: NCT06536842
Title: Postoperative Outcomes Following Primary Lumbar Fusion in Patients With and Without a Drain: A Prospective Randomized Control Trial
Brief Title: Wound Drain After Lumbar Fusion Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-2934CKEP
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Lumbar Fusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Postoperative Drain Group (Active Comparator): Participants will undergo their primary lumbar fusion spine surgery as planned and will have a drain placed postoperatively
  Interventions: Other: Postoperative Drain Placement
- Group 2: No Postoperative Drain Group (Active Comparator): Participants will undergo their primary lumbar fusion spine surgery as planned and will not have a drain placed postoperatively
  Interventions: Other: No Postoperative Drain Placement

INTERVENTIONS:
Other: Postoperative Drain Placement — These drains will be placed with the intention to decrease the incidence of postoperative hematoma
  Arms: Group 1: Postoperative Drain Group
Other: No Postoperative Drain Placement — Participant will undergo lumbar spine fusion surgery and will not receive a postoperative drain
  Arms: Group 2: No Postoperative Drain Group

SUMMARY:
Postoperative drain placement is often used following spine surgery. These drains are placed with the intention to decrease the incidence of postoperative hematoma and its associated complications including wound complications, infections and neurologic compression.

The use of drains, however, are not without its disadvantages including the risk of retrograde infection, increased postoperative blood loss, increased length of stay and increased hospital costs. The purpose of this study is to evaluate the postoperative outcomes and complications in patients undergoing primary lumbar fusion with and without a postoperative drain

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Undergoing primary lumbar fusion or decompression and fusion for 1-2 levels
* Surgery indicated for lumbar degenerative disease

Exclusion Criteria:

* Undergoing revision surgery
* Surgery indicated for infection
* Intraoperative dural tear
* Surgery requiring intraoperative transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative complications | 1 year
  Incidence of postoperative complications will be measured but recording the number of emergency department visits

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States